CLINICAL TRIAL: NCT00107393
Title: Phase II Study of Trastuzumab (Herceptin) and Capecitabine (Xeloda) in Women With Taxanes and Anthracyclines Refractory Metastatic Breast Cancer and HER2 Over-Expression
Brief Title: Trastuzumab and Capecitabine in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tohoku University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: TUGSM-UHA-BC03-01; CDR0000380787 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2006-10

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Capecitabine

INTERVENTIONS:
Biological: trastuzumab
Drug: capecitabine

SUMMARY:
RATIONALE: Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving trastuzumab together with capecitabine may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving trastuzumab together with capecitabine works in treating women with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the median survival time and 2-year survival rate in women with taxane- and anthracycline-refractory HER2/neu-overexpressing metastatic breast cancer treated with trastuzumab (Herceptin®) and capecitabine.

Secondary

* Determine the progression-free survival of patients treated with this regimen.
* Determine the response rate in patients treated with this regimen.
* Determine the clinical benefit rate of this regimen in these patients.
* Determine the safety profile of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to prior treatment with trastuzumab (Herceptin®) (yes vs no), HER2/neu status (3+ by immunohistochemistry vs positive by fluorescence in situ hybridization), and class of refractory disease (primary vs secondary vs treatment discontinuation due to adverse events).

Patients receive oral capecitabine once daily on days 1-21 and trastuzumab IV on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for up to 2 years.

PROJECTED ACCRUAL: A total of 75 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Metastatic disease

    * Patients with only bone metastases are not eligible
* Refractory disease, defined as disease progression, drug-related adverse reaction, or disease relapse during or within 12 months after completion of paclitaxel or docetaxel AND doxorubicin or epirubicin administered in the neoadjuvant, adjuvant, or metastatic setting

  * Total neoadjuvant or adjuvant taxane dose > 700 mg/m^2 for paclitaxel or > 240 mg/m^2 for docetaxel
  * Total taxane dose > 350 mg/m^2 for paclitaxel or > 120 mg/m^2 for docetaxel in the metastatic setting
  * Total neoadjuvant or adjuvant anthracycline dose > 240 mg/m^2 for doxorubicin or epirubicin
  * Total anthracycline dose > 120 mg/m^2 for doxorubicin or epirubicin in the metastatic setting
* HER2/neu overexpression

  * 3+ by immunohistochemistry or positive by fluorescence in situ hybridization
* No symptomatic brain metastases
* No pleural or pericardial effusion or ascites
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 20 to 75

Sex

* Female

Menopausal status

* Not specified

Performance status

* ECOG 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL

Hepatic

* SGOT or SGPT ≤ 2.0 times upper limit of normal (ULN) (< 3.0 times ULN for patients with liver metastases)
* Alkaline phosphatase ≤ 2.5 times ULN
* Bilirubin ≤ 1.5 mg/dL

Renal

* Creatinine ≤ 1.2 mg/dL

Cardiovascular

* LVEF > 50%

Pulmonary

* No interstitial pneumonia with pulmonary fibrosis

Other

* No history of hypersensitivity reactions
* No serious, uncontrolled infection
* No other malignancy
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior trastuzumab (Herceptin®) for metastatic disease allowed

Chemotherapy

* See Disease Characteristics
* No prior capecitabine
* At least 2 weeks since prior antimetabolites for metastatic disease
* At least 4 weeks since prior alkylating agents, carcinostatic antibiotics, or other carcinostatic agents

Endocrine therapy

* At least 4 weeks since prior goserelin or leuprolide for metastatic disease
* At least 2 weeks since prior oral endocrine agents for metastatic disease
* No concurrent endocrine therapy

Radiotherapy

* No prior radiotherapy to target lesions
* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy, including radiotherapy for brain metastases

Surgery

* Not specified

Other

* Concurrent bisphosphonates for bone metastases allowed

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2003-06; Primary Completion 2008-05 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Median survival and 2-year survival rate as measured by the Kaplan-Meier method 2 years after completion of study treatment

SECONDARY OUTCOMES:
Progression-free survival
Response rate
Clinical benefit rate as measured by Kaplan-Meier method 2 years after completion of study treatment
Safety profile as measured by the Kaplan-Meier method 2 years after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Noriaki Ohuchi, MD, Study Chair — Tohoku University
Locations (10):
- Japan (10):
  - Kitakyushu Municipal Medical Center, Fukuoka
  - Hiroshima University Hospital, Hiroshima
  - Hokkaido Cancer Center, Hokkaido
  - Saint Marianna University School of Medicine, Kanagawa
  - National Hospital Organization - Osaka National Hospital, Osaka
  - Osaka Kosei Nenkin Hospital, Osaka
  - Osaka University Graduate School of Medicine, Osaka
  - Tohoku University Graduate School of Medicine, Sendai
  - St. Luke's International Hospital, Tokyo
  - Sakata Municipal Hospital, Yamagata

REFERENCES:
- [Result] Ishida T, Kiba T, Takeda M, Matsuyama K, Teramukai S, Ishiwata R, Masuda N, Takatsuka Y, Noguchi S, Ishioka C, Fukushima M, Ohuchi N. Phase II study of capecitabine and trastuzumab combination chemotherapy in patients with HER2 overexpressing metastatic breast cancers resistant to both anthracyclines and taxanes. Cancer Chemother Pharmacol. 2009 Jul;64(2):361-9. doi: 10.1007/s00280-008-0882-8. Epub 2008 Dec 12. PMID 19082596